CLINICAL TRIAL: NCT00877370
Title: Pharmacokinetics of Invanz® (Ertapenem) in Critically Ill Patients Receiving Continuous Venovenous Hemodialysis
Brief Title: Pharmacokinetics of Ertapenem in Continuous Venovenous Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Bruce A. Mueller, Professor of Pharmacy, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HUM00022460
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-08

CONDITIONS: Acute Kidney Failure
Keywords: ertapenem; continuous hemodialysis; pharmacokinetics
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ertapenem (Experimental): subjects will receive ertapenem while receiving CVVHD
  Interventions: Drug: ertapenem

INTERVENTIONS:
Drug: ertapenem — One gram ertapenem will be infused intravenously in subjects receiving continuous hemodialysis (CVVHD). Pharmacokinetic sampling in this study will occur with the first dose of ertapenem. While on CVVHD, enrolled subjects will receive ertapenem 1 g intravenously administered over 30 minutes. Two blood samples (5 mL each) will be collected from the arterial (pre-diafilter) port of the CVVHD tubing at time 0 (baseline), ½ hour (end of infusion), 1, 1½, 2, 3, 6, 12, and 24 hours. Effluent (5 mL) will also be collected at these predefined time points from the effluent port of the CVVHD tubing. If ertapenem is discontinued after the first dose then additional samples will be collected at 36 and 48 hours, otherwise ertapenem will be administered as soon as the 24 hour sample is obtained.
  Other Names: Invanz

SUMMARY:
Critically ill patients in the intensive care unit often receive continuous hemodialysis to treat their kidney failure. Ertapenem is an antibiotic often used in these patients. Continuous dialysis may remove ertapenem, putting patients at risk for inappropriate treatment of their infection. This study will determine how much ertapenem is removed by continuous hemodialysis.

DETAILED DESCRIPTION:
Subjects receiving CVVHD will receive a one gram dose of ertapenem. Serial blood samples over 24 hours will be taken to assess the ertapenem blood concentrations over time. Spent dialysate and urine samples (if any) will also be measured for ertapenem content to determine how much drug is removed by CVVHD and kidneys. A pharmacokinetic evaluation will be made to determine what is the most appropriate dose for this drug in patients receiving CVVHD to achieve pharmacokinetic and pharmacodynamic goals.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in ICU
* Receiving Continuous hemodialysis
* Prescribed ertapenem
* Informed consent granted

Exclusion Criteria:

* < 18 years of age
* Allergy to ertapenem or other carbapenem antibiotic
* Severe, life-threatening reaction to penicillin or cephalosporins
* Patients experiencing or with history of CNS disorders (eg: seizure, stroke)
* Patients experiencing CNS infection
* Inability to complete 24 hours of CVVHD
* Concurrent use of other extracorporeal therapies such as extracorporeal membrane oxygenation, plasmapheresis or intermittent hemodialysis
* Inability to obtain informed consent
* Pregnant and/or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Mueller, Pharm.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan University Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Eyler RF, Vilay AM, Nader AM, Heung M, Pleva M, Sowinski KM, DePestel DD, Sorgel F, Kinzig M, Mueller BA. Pharmacokinetics of ertapenem in critically ill patients receiving continuous venovenous hemodialysis or hemodiafiltration. Antimicrob Agents Chemother. 2014;58(3):1320-6. doi: 10.1128/AAC.02090-12. Epub 2013 Dec 9. PMID 24323468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were consented and enrolled between April 2009 and March 2011. All subjects were patients receiving care in an intensive care unit at University of Michigan Health System.
Pre-assignment Details: All patients that qualified for the study were approached. All subjects that gave their consent were enrolled.
Groups:
- Ertapenem: Subjects will receive ertapenem while receiving CVVHD
  ertapenem : One gram ertapenem will be infused intravenously in subjects receiving continuous hemodialysis (CVVHD). Pharmacokinetic sampling in this study will occur with the first dose of ertapenem. While on CVVHD, enrolled subjects will receive ertapenem 1 g intravenously administered over 30 minutes. Two blood samples (5 mL each) will be collected from the arterial (pre-diafilter) port of the CVVHD tubing at time 0 (baseline), ½ hour (end of infusion), 1, 1½, 2, 3, 6, 12, and 24 hours. Effluent (5 mL) will also be collected at these predefined time points from the effluent port of the CVVHD tubing. If ertapenem is discontinued after the first dose then additional samples will be collected at 36 and 48 hours, otherwise ertapenem will be administered as soon as the 24 hour sample is obtained.
Period: Overall Study
Arm/Group | Ertapenem
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ertapenem
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 62 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Ertapenem Transmembrane Clearance by Continuous Hemodialysis.
Time Frame: 24 hours after receiving first 1 gram dose
Population: All participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Ertapenem
Number analyzed (Participants) | 8
mL/min | 10.4 (4.2)

ADVERSE EVENTS:
Arm/Group | Ertapenem
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No